CLINICAL TRIAL: NCT01093287
Title: Predictors for Responsiveness to Corticosteroid in Patients With Early Acute Respiratory Distress Syndrome
Status: Terminated | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gee Young Suh, Professor, Samsung Medical Center
Other Study IDs: 2009-08-075
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In a recent multicenter randomized controlled trial, prolonged administration of low-dose methylprednisolone (1mg/kg/day) initiated in early acute respiratory distress syndrome was associated with earlier resolution of pulmonary and extrapulmonary organ dysfunction and reduction in duration of mechanical ventilation and intensive care unit stay. However, glucocorticoids may induce serious adverse events and these adverse events might compensate the positive effect of prolonged methylprednisolone infusion and discourage physicians from treating acute respiratory distress syndrome patients with glucocorticoids. Early prediction of responsiveness to prolonged methylprednisolone infusion would be help to decide whether to continue or not prolonged methylprednisolone infusion and this could reduce the drug related adverse events. We project to evaluate the predictors of responsiveness to prolonged methylprednisolone infusion in early acute respiratory distress syndrome .

ELIGIBILITY:
Inclusion Criteria:

* AECC definition of acute respiratory distress syndrome
* Early acute respiratory distress syndrome (within 72 h of diagnosis)
* PF ratio < 200 at PEEP ≥ 8 cmH2O

Exclusion Criteria:

* Imminent death
* Contraindication to corticosteroid treatment
* Already on more than 0.5 mg/kg of methylprednisolone or its equivalent
* Evidence of uncontrolled infection
* Refusal of managing physician to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the American European Consensus definition of acute respiratory distress syndrome will be included, regardless of etiology of respiratory failure.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jeon K, Chung CR, Yang JH, Park CM, Suh GY. Predictors of response to corticosteroid treatment in patients with early acute respiratory distress syndrome: results of a pilot study. Yonsei Med J. 2015 Jan;56(1):287-91. doi: 10.3349/ymj.2015.56.1.287. PMID 25510776